CLINICAL TRIAL: NCT04713124
Title: Ready2Change-Methamphetmine (R2C-M): A Randomised Controlled Trial of a Telephone-delivered Intervention to Reduce Methamphetamine Use
Brief Title: A Telephone-delievered Intervention to Reduce Methamphetamine Use
Acronym: R2C-M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turning Point (Other)
Collaborators: Eastern Health (Other); Monash University (Other); Deakin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E20/011/61428
Record Dates: First submitted 2021-01-11; First posted 2021-01-19 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Methamphetamine Use Disorder

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R2C-M intervention (Experimental): R2C-M telephone intervention - Six approximately weekly sessions of R2C-M telephone-delivered intervention (50 minutes in duration), delivered by the same R2C-M Counsellor each session (a qualified clinical psychologist trained in the R2C protocol by the developer, Dr Kate Hall). Call duration will be recorded. Sessions will be digitally recorded, and an independent researcher will randomly select and rate fidelity of intervention sessions for 20% of participants.
  R2C-M workbooks - Two workbooks to facilitate counsellor-delivered exercises within sessions, and between-session practice, will be mailed/emailed to participants.
  Self-help booklet - (as in control group) R2C-M participants will also receive a booklet of information and self-help strategies for methamphetamine use problems.
  Interventions: Behavioral: R2C-M; Other: Self-help booklet
- Control (Active Comparator): Self-help booklet - Control participants will receive (by mail/email) a booklet of information and self-help strategies for methamphetamine use problems.
  Telephone check-ins + information on further support - (to control for frequency of contact across treatment arms) Participants in this group will receive 6 telephone calls from the research team (lasting maximum 5 minutes, call duration will be recorded). During these calls, participants will be asked about their use of the booklet. Whenever required, the researcher will provide participants with information on further support (e.g. DirectLine or other state/territory AOD helpline for advice or referral).
  Interventions: Other: Self-help booklet

INTERVENTIONS:
Behavioral: R2C-M — R2C-M comprises 12 modules addressing core practice elements and skills from evidence-based cognitive and behavioural interventions. Modules include: (i) self-monitoring, goal setting and behaviour change skills; (ii) identification of strengths and motivational enhancement; (iii) relapse prevention; (iv) psychoeducation and harm reduction; (v) emotion regulation skills; (vi) anger management skills; (vii) urges and cravings management skills; (viii) sleep hygiene skills; (ix) mindfulness skills; (x) interpersonal skills; (xi) anxiety management skills; (xii) depressed mood management skills. The R2C-M workbooks contain psychoeducation and intervention exercises, to facilitate counsellor-delivered exercises within sessions, and between-session practice.
  Arms: R2C-M intervention
Other: Self-help booklet — A booklet of information and self-help strategies for methamphetamine use problems.

SUMMARY:
Australia has one of the highest rates of methamphetamine use in the world; however, uptake of face-to-face psychological treatment remains extremely low due to numerous individual (e.g. stigma, shame) and structural (e.g. service availability, geography) barriers to accessing care. Addressing these barriers through the provision of alternative treatment delivery models is imperative, particularly as effective and earlier intervention is likely to reduce the need for more costly and intensive treatment resulting from escalating methamphetamine use.

In this project, the investigators will conduct the first double-blind, parallel-group, randomised controlled trial (RCT) examining the effectiveness of the structured telephone-delivered intervention, Ready2Change (R2C), among participants with methamphetamine use problems (R2C-M). Cost effectiveness of R2C-M will also be investigated. Factors influencing program implementation will be evaluated to inform the scalability of this intervention for practice nationally, and for replication internationally.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years
* Mild or moderate methamphetamine use disorder (DSM-5 diagnosis confirmed at baseline assessment using the Structured Clinical Interview for DSM-5 Disorders - Research Version, SCID-5-RV)
* Used methamphetamine on at least two occasions in the past month
* Seeking to reduce methamphetamine use
* Able to provide informed consent, and comply with the requirements of the treatment protocol
* Willing to provide the contact details of their general practitioner or other treating physician, for follow-up
* English as a first language or fluent
* Educated to high school level (literacy)
* Regular access to a telephone
* Postal/email address to receive intervention materials

Exclusion Criteria:

* Currently receiving treatment for substance use disorder (e.g. medically supervised detoxification, residential rehabilitation, drug counselling, pharmacotherapy - this criterion applies only at trial enrolment, and does not preclude the participant from entering treatment/receiving usual care during the trial)
* Requiring acute care for severe substance use disorder (DSM-5 diagnosis confirmed at baseline using the SCID-5-RV, with oversight from the Principal Investigator or Study Clinician)
* Requiring acute care for active suicidality or unstable psychiatric condition
* A diagnosed primary psychotic disorder (schizophrenia, schizoaffective disorder, bipolar disorder)
* Pregnancy
* Hearing impairment that would prohibit participation in telephone intervention / follow-up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Methamphetamine problem severity | 3-months post-randomisation
  Change in methamphetamine problem severity (Drug Use Disorders Identification Test; DUDIT)

SECONDARY OUTCOMES:
Methamphetamine problem severity | 6- and 12-months post-randomisation
  Change in methamphetamine problem severity (DUDIT)
Number of methamphetamine use days | 6 weeks, and 3-, 6- and 12-months post-randomisation
  Change in number of methamphetamine use days (Timeline Followback; TLFB)
Amount of methamphetamine used | 6 weeks, and 3-, 6- and 12-months post-randomisation
  Change in amount of methamphetamine used (TLFB)
Number of DSM-5 methamphetamine use disorder criteria met | 3-, 6- and 12-months post-randomisation
  Change in the number of DSM-5 methamphetamine use disorder criteria met (Structured Clinical Interview for DSM-5 Disorders - Research Version; SCID-5-RV)
Methamphetamine craving | 6 weeks, and 3-, 6- and 12-months post-randomisation
  Change in craving for methamphetamine (Craving Experience Questionnaire; CEQ)
Psychological functioning | 6 weeks, and 3-, 6- and 12-months post-randomisation
  Change in psychological functioning (Depression Anxiety and Stress Scale; DASS-12)
Psychotic-like experiences | 6 weeks, and 3-, 6- and 12-months post-randomisation
  Change in psychotic-like experiences (Community Assessment of Psychic Experiences 15, CAPE15)
Quality of life | 6 weeks, and 3-, 6- and 12-months post-randomisation
  Change in quality of life (EUROHIS-QOL single item)
Days of other drug use | 6 weeks, and 3-, 6- and 12-months post-randomisation
  Change in days of other drug use (TLFB)
Cost-effectiveness - QALYs | Over 12 months
  Difference in quality-adjusted life years (QALYs) (abridged version of the 5-level EQ-5D version, EQ-5D-5L+)
Cost-effectiveness - health care costs | Over 12 months
  Difference in health care costs (3Mg Health-care Resource Use Questionnaire)
Cost-effectiveness - work-related losses | Over 12 months
  Difference in work-related losses (World Health Organization Health and Performance Questionnaire Clinical Trials Version; WHO HPQ28-Day)
Adverse events | Up to 6 weeks post-randomisation
  Occurrence of adverse events (AEs) and significant adverse events (SAEs)

OTHER OUTCOMES:
Program evaluation | Through study completion, approximately 28 months
  Mixed-methods program evaluation (Glasgow et al.'s RE-AIM framework)

CONTACTS AND LOCATIONS:
Overall Officials: Dan I Lubman, Principal Investigator — Turning Point, Eastern Health; Monash University
Locations (1):
- Turning Point, Richmond, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
No Ethics approval to seek patient permission to share data outside this study, other than for related projects conducted by the research team.

REFERENCES:
- [Derived] Lubman DI, Manning V, Arunogiri S, Hall K, Reynolds J, Stragalinos P, Petukhova R, Gerhard R, Tyler J, Bough A, Harris A, Grigg J. A structured, telephone-delivered intervention to reduce methamphetamine use: study protocol for a parallel-group randomised controlled trial. Trials. 2023 Mar 29;24(1):235. doi: 10.1186/s13063-023-07172-9. PMID 36991490

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT04713124/SAP_000.pdf